CLINICAL TRIAL: NCT00787397
Title: Sleep, Mood, and Behavior Study:Transdisciplinary Studies of CBT for Anxiety in Youth
Brief Title: Sleep, Mood, and Behavior Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Neal Ryan, Joaquim Puig-Antich Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO08010426; P50MH080215-01A1 (NIH)
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Difficulties in Pediatric Anxiety Disorder; Generalized Anxiety Disorder; Separation Anxiety Disorder; Social Phobia
Keywords: Sleep difficulties in pediatric anxiety disorder; Neural correlates of pediatric anxiety disorder; Social correlates of pediatric anxiety disorder; Generalized Anxiety Disorder in pediatric populations; Separation Anxiety Disorder in pediatric populations; Social Phobia in pediatric populations
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1. Cognitive Behavioral Therapy-Sleep (Experimental): Cognitive Behavioral Therapy-Sleep
  Interventions: Behavioral: Cognitive Behavioral Therapy-Sleep

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Sleep — Cognitive Behavioral Therapy: 6 sessions of CBT

SUMMARY:
The purpose of this study is to assess whether improving sleep in children and adolescents with anxiety disorder will further enhance affective, clinical, and social functioning.

DETAILED DESCRIPTION:
This study is one of two interlinking protocols developed to investigate neural, affective, behavioral and social predictors of improvement as a critical next step in advancing the understanding of processes involved in the treatment response of anxiety disorders in youth. This protocol will offer a six to eight session sleep intervention (Sleeping Tigers)children ages 9-13 who currently have a DSM-IV anxiety disorder and who endorse some level of impairment in their ability to sleep. Participants will have completed a 16 session intervention for anxiety (IRB submission, Child Anxiety Treatment Study CATS). We hope to assess whether improving sleep will further enhance affective, clinical, and social functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of DSM-IV diagnosis of Generalized Anxiety Disorder (GAD), Separation Anxiety Disorder (SAD), and Social Phobia (SP)
2. Previous enrollment Cognitive Behavioral Therapy arm in ClinicalTrials.gov Identifier: NCT00774150 study, entitled, " Transdisciplinary Studies of CBT for Anxiety in Youth: Child Anxiety Treatment Study (CATS)"
3. The child/adolescent must have a "sleep problem" defined as: difficulties at least 3 times within a 2-week period in one or more of the following domains:

   * difficulties going to sleep
   * difficulties waking during the night
   * difficulties getting up on time for school because of tiredness/sleepiness
   * daytime tiredness and/or irritability that the child or parent attributed to insufficient sleep
   * erratic sleep-wake schedules

Exclusion Criteria:

1. IQ below 70 as assessed by the Wechsler Abbreviated Scale of Intelligence (WASI).
2. Requires current ongoing treatment with psychoactive medications including anxiolytics and antidepressants.
3. Acutely suicidal or at risk for harm to self or others.
4. Any motor impairments or eye-hand coordination problems
5. Sleep disorder or parasomnia.
6. Taking any medication that might interfere with sleep.
7. Has a medical problem that might interfere with sleep.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evidence of sleep therapy effects on anxiety symptoms are established by assessments of clinical status, symptoms, affective style, sleep,parent-child interactions using rating scales, self-report measures, and behavioral observations. | 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Ryan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States